CLINICAL TRIAL: NCT06280456
Title: The Efficacy of Intra-articular Tranexamic Acid Injection With Different Drainage Clamping Time in Postoperative Bleeding and Pain After Arthroscopic Anterior Cruciate Ligament Reconstruction
Brief Title: Tranexamic Acid Injection With Different Drainage Clamping Time After Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-09-017A
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-09

CONDITIONS: Anterior Cruciate Ligament Reconstruction; Tranexamic Acid; Hemarthrosis, Knee
MeSH Terms: conditions — Hemarthrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic Acid 4-hour group (Experimental): 10 mL of TXA (100 mg/mL) was injected into the joint at the end of the index operation and the drain was clamped for 4 hours.
  Interventions: Drug: Tranexamic Acid Powder
- Tranexamic Acid 8-hour group (Experimental): 10 mL of TXA (100 mg/mL) was injected into the joint at the end of the index operation and the drain was clamped for 8 hours.
  Interventions: Drug: Tranexamic Acid Powder

INTERVENTIONS:
Drug: Tranexamic Acid Powder — 10 mL of Tranexamic Acid(100 mg/mL) was injected into the joint at the end of the operation with different drainage clamping time.
  Other Names: Daiichi Sankyo

SUMMARY:
Post-anterior cruciate ligament reconstruction (ACLR) hemarthrosis may result in increased pain thus delaying postoperative rehabilitation, which may eventually lead to arthrofibrosis and a functional deficit. Many antifibrinolytic agents, including tranexamic acid (TXA), have been used in orthopedic surgeries to reduce postoperative bleeding. Moreover, TXA was proved effective to reduced the events of hemarthrosis and increased the post-operative functional outcomes of the patients in several studies. The purpose of this study is to evaluate the efficacy of intra-articular injection of TXA with different drainage clamping time in patients receiving arthroscopic ACLRs. Patients were randomized into four groups. An intra-articular suction drain was placed recorded 24 h postoperatively. Group 1 patients(TXA 4hr group) received the index procedures with a 10 mL intra-articular injection of TXA and following drainage clamped 4 hours. Group 2 patients(TXA 8hr group) received the index procedures with a 10 mL intra-articular injection of TXA and following drainage clamped 8 hours. Clinical evaluations using an IKDC functional score and a Visual Analogue Scale (VAS) pain score were performed during admission, at postoperative day 3 and week 4.

DETAILED DESCRIPTION:
Surgical technique All patients participating in this study received surgery by the same surgeon (H.L.M.) with spinal anesthesia. Pneumatic tourniquet was routinely utilized during the procedure. A 3-cm incision was made over the medial proximal tibia to harvest the semitendinosus and gracilis tendons from the distal insertion. The tendons were quadrupled and whipstitched with No. 2 and No. 5 Ethibond sutures (Ethicon, Somerville, NJ) as previously described.12 The folded tendons' diameters were measured using sizing cylinders with 0.5 mm incremental changes in size. The femoral sockets were created by drilling from the insertion site at the lateral femoral condyle through the anteromedial portal. The tibial tunnel was drilled with an Acufex guide (Smith & Nephew, Andover, MA). The diameters of the sockets were matched to the size of the folded graft. The grafts were fixed with bioscrews (BioRCI-HA; Smith & Nephew) at the femoral site and at the tibial site with the knee flexed at 30°. The screw and tunnel sizes were identical. Following the procedure, a Hemovac suction drain (Zimmer, Warsaw, IN) was placed at the superior-lateral aspect of the joint. Additionally, in the TXA group, 10 mL of TXA solution (100 mg/mL; Daiichi Sankyo, Tokyo, Japan) was injected into the joint, and all closed suction drains were clamped for 4, or 8 hours based on the grouping results.

Clinical evaluation Postoperative drainage output is the primary outcome of this study. The drain tubes were routinely removed postoperatively once the volume of drainage decreased, of which the total volume was recorded. The secondary outcomes included visual analog scale (VAS) and International Knee Documentation Committee (IKDC) functional score. The former was documented immediately after patients were transferred back to the ward from the post-anesthesia recovery room, on day 3 and at week 4 after surgery. Besides, the maximum of postoperative VAS score during admission was also documented. IKDC functional score was a subjective questionnaire including three categories with symptoms, athletic activity, and knee function. Higher score indicated better function with highest score of 10 and lowest of 0. All the objective measurements followed at postoperative 4 week were evaluated by an independent observer who was blinded to this study at the outpatient clinic.

Statical analysis The power calculation was calculated using the G*Power software (version 3.1; Heinrich-Heine-Universität Düsseldorf, Düsseldorf, Germany). The volume of drainage between groups from our previous study was used as the primary variable. With a power of 0.8 and a significance level of .05, a total of 49 patients were required for each group. Oversampling of patients in each group was performed due to potential withdrawals and losses to follow-up. All data are expressed as mean and 95% confidence interval or standard deviation. The amounts of drainage and the functional scores were compared among four groups with Analysis of Variance(ANOVA) with post-hoc Tukey Honestly Significant Difference test. All statistical analyses were conducted using SPSS software (version 22.0, IBM, Armonk, NY). Differences were considered significant at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Receiving arthroscopic anterior cruciate ligament reconstruction with autologous hamstring grafts

Exclusion Criteria:

* previous knee procedure on the same side
* renal diseases
* coagulation disorder
* refusal of participation in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
The volume of drainage | 1 day (Total volume was recorded once the drain tube removed)
  hemarthrosis

SECONDARY OUTCOMES:
Visual analog scale (VAS) | Immediately when back to the ward, maximum during admission, postoperative day 3 and week 4
  Scale 0 to 10.
International Knee Documentation Committee (IKDC) functional score | Evaluated 4 weeks post-surgery.
  Score 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: En-Rung Chiang, Study Chair — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan